ACE-MY-001

Statistical Analysis Plan

Version 2.0 dated: 20 September 2018

**Protocol Number: ACE-MY-001** 

Protocol Title: An Open-label, Phase 1b Study of ACP-196 in Subjects with

**Multiple Myeloma** 

Version: 2.0

Version date: 20 September 2018

The undersigned have reviewed this plan and find it to be consistent with the requirements of the protocol as it applies to their respective areas

Prepared by

Associate Director, Biostatistics



## **CONFIDENTIAL**

This document (and all copies thereof) is the property of Acerta Pharma and contains valuable trade secrets and confidential information, including proprietary technical and business information. By accepting this document, you agree that the Confidential Information contained herein will not be disclosed to others without prior written authorization from Acerta Pharma and shall only be used for the purposes intended by the document.

# **Statistical Analysis Plan**

An Open-label, Phase 1b Study of ACP-196 in Subjects with Multiple Myeloma

**Protocol Number: ACE-MY-001** 

Version: Date: Study Statistician: Version 2.0 20 September, 2018

Acerta Pharma 

## **TABLE OF CONTENTS**

| Tabl | le of Contents | 2 |
|---|---|---|
| Tabl | ole of Abbreviations | 4 |
| 1. | INTRODUCTION | 5 |
| 2. | OBJECTIVES | 5 |
| 3. | STUDY OVERVIEW 3.1 Study Design | 6 |
| 4. | STUDY ENDPOINTS | 7<br>7 |
| 5. | HYPOTHESES AND MULTIPLICITY | 7 |
| 6. | ANALYSIS SETS | 8 |
| 7. | INTERIM ANSLYSIS AND EARLY STOPPING GUIDELINES | 8 |
| 8. | FINAL ANALYSIS AND CLINICAL STUDY REPORT | 8 |
| 9. | MISSING VALUES | 8 |
| 10. | STATISTICAL METHODS OF ANALYSIS 10.1 General Principles 10.2 Subject Disposition 10.3 Important Protocol Deviations 10.4 Baseline Data 10.4.1 Demographics 10.4.2 Baseline Characteristics 10.4.3 Baseline Disease Characteristics | 9<br>9<br>9<br>10 |
| | 10.5 Treatment and Medications | |

| | 10.5.2 Prior and Concomitant Medications Received for Indications Other Than MM | 11 |
|---|---|---|
| | 10.5.3 Exposure to Study Drugs | .12 |
| | 10.6 Analyses of Safety Endpoints | .12 |
| | 10.6.1 Adverse Events of Clinical Interest | .13 |
| | 10.6.2 Laboratory Abnormality | .14 |
| | 10.6.3 Vital Signs | .15 |
| | 10.6.4 ECOG Performance Score | .15 |
| | 10.6.5 Electrocardiogram | .16 |
| | 10.7 Analyses of Efficacy Endpoints | .16 |
| | 10.7.1 Definitions | .16 |
| | 10.7.2 Analysis Methods | .17 |
| 11. | DISEASE BIOMARKERS | .17 |
| 12. | CHANGES FROM PROTOCOL-SPECIFIED ANALYSES | .17 |
| 13. | LITERATURE CITATIONS / REFERENCES | .18 |
| 14. | APPENDICES | 19 |
| | 14.1 Definitions | |
| | 14.1.1 Study Day | .19 |
| | 14.2 Imputation Rules | |
| | 14.2.1 Partial or Missing Dates | .19 |
| | 14.3 Censoring Rules for Duration of Response and Progression-Free Survival. | .20 |
| | 14.4 Events of Clinical Interest | .20 |

#### **TABLE OF ABBREVIATIONS**

AE(s) adverse event(s)
Bid twice per day

CBR clinical benefit rate
CR complete response
CSR clinical study report

CTCAE Common Terminology Criteria for Adverse Events

DCR disease control rate
DOR duration of response

ECOG Eastern Cooperative Oncology Group
Ex-US Excluding United States of America

lg immunoglobulin

IRC independent review committee
IPD important protocol deviation
ISS International Staging System

MedDRA Medical Dictionary for Regulatory Activities

MM multiple myeloma
MR minimal response

NCI National Cancer Institute

PD pharmacodynamics

PFS progression-free survival

PK pharmacokinetics
PR partial response
PT preferred term

SAE(s) serious adverse event(s) SAP statistical analysis plan

sCR stringent complete response

SD stable disease

TEAE(s) treatment-emergent adverse events

VGPR very good partial response WHO World Health Organization

#### 1. INTRODUCTION

The purpose of this statistical analysis plan (SAP) is to provide details of the safety and efficacy analyses that have been outlined within Protocol Amendment 2 for Study ACE-MY-001, which is entitled "An Open-label, Phase 1b Study of ACP-196 in Subjects with Multiple Myeloma" dated January 13, 2016. The original SAP based on same protocol was for interim safety clinical study report (CSR) to support the new drug application (NDA) in relapsed and refractory mantle cell lymphoma. This SAP is updated to include efficacy analysis. Any change to the planned analyses described in the final SAP will be documented in the clinical study report (CSR).

Separate reports will be generated for pharmacokinetic (PK) and pharmacodynamic (PD) data.

From here on, acalabrutinib (generic name for formerly ACP-196) will be used in place of ACP-196 in this document.

#### 2. OBJECTIVES

## 2.1 **Primary Objective**

 To characterize the safety profile of acalabrutinib with and without dexamethasone in subjects with relapsed or refractory (R/R) multiple myeloma (MM).

## 2.2 Secondary Objectives

- To characterize the PK profile of acalabrutinib with and without dexamethasone and the PK profile of dexamethasone with concomitant acalabrutinib administration
- To evaluate the PD effects of acalabrutinib with and without dexamethasone
- To evaluate the activity of acalabrutinib with and without dexamethasone as measured by overall response rate (ORR), duration of response (DOR), clinical benefit rate, disease control rate, and progression-free survival (PFS).
- To explore the relationship between biological markers in MM cells and response to therapy

#### STUDY OVERVIEW

## 3.1 Study Design

This study is a multicenter, open-label, randomized, parallel-group study to be conducted at approximately 20 sites in 2 countries (United Kingdom and United States). Forty subjects are planned to be randomized 1:1 into the following 2 cohorts to receive acalabrutinib, with or without dexamethasone:

- Cohort 1 (acalabrutinib monotherapy): acalabrutinib 100 mg bid continuously
- Cohort 2 (acalabrutinib + dexamethasone): acalabrutinib 100 mg bid continuously and 40 mg dexamethasone once weekly

Due to limited evidence of efficacy of acalabrutinib monotherapy in R/R MM subjects in this study, in a memo dated March 15, 2016 to all study sites, the enrollment was discontinued immediately and subjects who were randomized to receive acalabrutinib monotherapy were permitted to crossover to receive acalabrutinib + dexamethasone treatment.

One cycle is defined as a 28-day study treatment period. Treatment may be continued until disease progression (PD) or an unacceptable drug-related toxicity occurs. All subjects who discontinue study drug will have a safety follow-up visit 30 (±7) days after the last dose of study drug unless they have started another cancer therapy within that timeframe.

All subjects will have hematology, serum chemistry, and urinalysis safety panels done at screening. Once dosing commences (Day 1), all subjects will be evaluated for safety, including serum chemistry, and hematology, once weekly for the first 4 weeks, every 2 weeks in Cycle 2 and monthly thereafter. PK/PD testing will be done in Cycle 1 and Cycle 2. The end of trial is defined as the point when the last subject on the study exits the study for any reason.

#### 3.2 Sample Size

The trial seeks to exclude an uninteresting ORR of ≤15% (i.e., the response rate that might be associated with single-agent dexamethasone therapy [Anderson 2013]) in favor a target response rate of ≥40%. Considering a sample size of 19 subjects per cohort, the power to detect the difference between a null hypothesis response rate of 15% and an alternative-hypothesis response rate of 40% with a 0.025 one-sided significance level is 69% using a one-group, exact binomial test. A sample size of 19 subjects per cohort

Acerta Pharma 

will also provide a 97.5% 1-sided confidence interval centered around an expected ORR of 40% that excludes an ORR of 18.6% as a lower bound.

#### 4. STUDY ENDPOINTS

#### 4.1 **Safety Endpoints**

The safety of acalabrutinib with and without dexamethasone will be characterized by the type, frequency, severity, and relationship to study drug(s) of any treatment-emergent adverse events (AEs) or incidence of abnormalities of laboratory tests; serious adverse events (SAEs); or AEs leading to dose modification/delay or discontinuation of study treatment.

#### 4.2 **Efficacy Endpoints**

Assessments of acalabrutinib efficacy in this study will be based on the criteria of standardized tumor response and disease progression for MM ([Rajkumar 2011] and [Blade 1998]).

- Overall response rate (ORR)
- Duration of response (DOR)
- Clinical benefit rate (CBR)
- Disease control rate (DCR) •
- Progression-free survival (PFS)

#### 4.3 Pharmacokinetic and Pharmacodynamic Parameters

Refer to separate reports for PK and PD parameters.

#### HYPOTHESES AND MULTIPLICITY 5.

No formal statistical hypotheses will be tested. The clinical hypotheses are that acalabrutinib monotherapy and acalabrutinib + dexamethasone is safety and effective in subjects with R/R MM.

#### 6. **ANALYSIS SETS**

#### 6.1 **All-Treated Population**

All-treated population is defined as all enrolled subjects who receive ≥ 1 dose of any study drug. All-treated population will be used for evaluating the safety and efficacy unless otherwise specified.

#### 6.2 Treatment Cohorts

Subjects are randomized with the ratio of 1:1 into 2 treatment cohorts to receive acalabrutinib, with or without dexamethasone:

- Cohort 1 (acalabrutinib monotherapy): acalabrutinib 100 mg bid continuously
- Cohort 2 (acalabrutinib + dexamethasone): acalabrutinib 100 mg bid continuously and 40 mg dexamethasone once weekly

#### 7. INTERIM ANALYSIS AND EARLY STOPPING GUIDELINES

No formal interim analysis will be conducted.

#### 8. FINAL ANALYSIS AND CLINICAL STUDY REPORT

The final analysis of primary and secondary efficacy endpoints will occur when last patient enrolled completes the end of Cycle 12, or withdraws for any reason and completes the 30-day follow-up visit, whichever occurs first. The CSR will be written based on the final analysis. The addendum of CSR will be written at the end of trial.

#### 9. MISSING VALUES

#### Missing Safety Data

Conservative imputation rules will be applied partial dates for AE onset and stop dates, start and end dates of concomitant medication, start date of subsequent anticancer therapy, date of initial diagnosis, and death date. The algorithm for the imputation in Appendices 14.2 will be used. If dates are completely missing, no imputation will be made. Missing safety data other than partial or missing dates will not be imputed.

#### 9.2 Missing Efficacy Data

The method of handing missing data and censoring data is described in the definition for the efficacy endpoints, mentioned at section 14.3.

#### 10. STATISTICAL METHODS OF ANALYSIS

#### 10.1 **General Principles**

Descriptive statistics will be used to summarize disposition, demographics, baseline characteristics, disease characteristics, prior anticancer therapy, concomitant medication, study drug administration, efficacy and safety outcomes. Descriptive summary of discrete data will be present the sample size and incidence as frequency and percentage. Descriptive summaries of continuous data will be present the sample size, group mean, standard deviation, median, and range.

Confidence intervals (CIs), when presented, will generally be constructed at the 95% level. For binomial variables, the exact method for CIs will be employed unless otherwise specified.

Calculation of time to event or duration of event (e.g., DOR) will be based on actual study day of event rather than nominal visit date.

## 10.2 Subject Disposition

Subjects are enrolled from 11 study sites of 2 countries. The number of subjects enrolled by region, country, and site will be presented. Subject disposition will be summarized for all enrolled subjects including the following information:

- Subject status on acalabrutinib
- Primary reasons for acalabrutinib discontinuation
- Subject status on the study
- Primary reasons for study discontinuation
- Time on the study

## 10.3 Important Protocol Deviations

Important Protocol Deviations (IPDs) categories are defined and managed by the study team during the IPD reviews throughout the study before database lock. These definitions of IPD categories, sub-category codes, and descriptions will be used during the course of the study. The final IPD list is used to produce the Summary of IPDs table.

#### 10.4 Baseline Data

Summaries of demographics and baseline characteristics will be presented for subjects in the All-treated population. For continuous variables, n, mean, standard deviation,

Acerta Pharma 

median, minimum, and maximum values will be provided. For categorical variables, the number and percentage of subjects in each category will be summarized.

## 10.4.1 Demographics

- Sex (Male, Female)
- Age (year, continuous)
- Age category (<65 versus ≥65 years)
- Ethnicity
  - Hispanic or Latino
  - Not Hispanic or Latino
  - Not Reported
- Race
  - American Indian or Alaska Native
  - Asian
  - Black or African American
  - Native Hawaiian or Other Pacific Islander
  - White
  - Other
  - Not Reported
- Country
  - Unites States
  - United Kingdom

## 10.4.2 Baseline Characteristics

- Eastern Cooperative Oncology Group (ECOG) performance score
  - 0 = fully active.
  - 1 = restricted in physically strenuous activity
  - 2 = incapable of any work activity
  - 3 = limited self-care
  - 4 = completely disabled
- Height (cm)
- Weight (kg)

#### 10.4.3 Baseline Disease Characteristics

• Time from initial diagnosis to first dose of acalabrutinib (months)

- Prior anticancer therapy regimens
  - Number of regimens (mean, standard deviation, median, minimum, maximum)
  - Number of subjects with regimens (1-3 regimens, >=4 regimens)
- Prior stem cell transplant
- MM stage by International Staging System (ISS) (stage I, II, III [Greipp 2005])
- MM subtypes
  - heavy chain subtypes
  - light chain subtypes
- Serum β2-microglobulin (<2.5, >=2.5 mg/L)
- Serum creatinine (<2, ≥ 2 mg/dL)
- Serum Hemoglobin (mean, standard deviation, median, min, max)
- Serum calcium (≤12, >12 g/dL)
- IgG (mean, median, min, max)
- IgA (mean, median, min, max)
- Bone marrow cellularity
  - Hypercellular
  - Normocellular
  - Hypocellular

## 10.5 **Treatment and Medications**

#### 10.5.1 **Prior Anticancer Therapies**

A prior anticancer therapy is defined as a systemic therapy subjects received, either as a single or combination therapy, for the treatment of MM with an end date occurring before the date of first dose of study treatment. Therapies given as a consolidation or for maintenance of a response or remission will not be considered as a separate regimen. The prior anticancer therapy regimens will be summarized.

# 10.5.2 Prior and Concomitant Medications Received for Indications Other Than MM

Concomitant therapy is defined as all medications used on or after the first dose of study drug, through the treatment phase, and through 30 days following the last dose of study drug. Data reported on concomitant medications CRF pages will be used. Medications

Acerta Pharma 

started prior to first dose of study drug will be consider as prior treatment. Using this definition, a medication can be classified as both prior and concomitant. The start date and end date will be based on the rules provided in Appendices 14.2.1. Medications with completely missing start and stop dates will be considered as both prior and concomitant medications. Prior and concomitant medications other than antineoplastic agents or other systemic therapies for MM after enrollment will be coded by the World Health Organization (WHO) Drug Dictionary and summarized by Anatomic Therapeutic Chemical Classification System (ATC) level 2 (therapeutic subgroup) and level 5 (preferred term/chemical ingredient).

#### 10.5.3 **Exposure to Study Drugs**

Separate analysis will be performed for acalabrutinib and dexamethasone. Descriptive statistics (n, mean, standard deviation, median, minimum and maximum values) will be used to summarize:

- Duration of exposure (the interval between first dose date and last dose date)
- Actual cumulative dose administered
- Average dose (the ratio of actual cumulative dose administered and Duration of exposure): daily dose for acalabrutinib and weekly dose for dexamethasone
- Relative dose intensities (the percentage of actual cumulative dose to the planned cumulative dose)

The reasons for acalabrutinib dose withholding and reduction will be summarized and presented as the number and percentage of subjects with non-missing data per category.

- Dose withholding of acalabrutinib is defined as missing dose for ≥ 7 consecutive days.
- Dose reduction defined as taking lower dose level (100 mg per day) for acalabrutinib for ≥ 3 consecutive days.

#### 10.6 **Analyses of Safety Endpoints**

Safety analyses will be performed on All-treated population by treatment cohort.

Analyses of adverse events (AEs) will be performed on treatment-emergent AE (TEAE) data, unless otherwise specified. TEAEs are defined as those events with onset or

Acerta Pharma  worsen date on or after the date of first dose of acalabrutinib, through the treatment phase to last dose of acalabrutinib, and within 30 days following the last dose of acalabrutinib, whichever is later. Common Terminology Criteria for Adverse Events (CTCAE) Version 4.03 or higher is used for AE grading.

Treatment-emergent AEs will be summarized in 3 groups: (1) acalabrutinib monotherapy, (2) acalabrutinib + dexamethasone, and (3) crossover from monotherapy to acalabrutinib + dexamethasone therapy. By this grouping method, AEs among subjects assigned to acalabrutinib monotherapy will be reported in group 1 when AEs occurred before crossover, and AEs occurred on/after crossover will be reported in group 3. Treatment-emergent AEs occurred on or after crossover will be summarized in the crossover group. Treatment-emergent AEs occurred before crossover will be summarized in the monotherapy group. All AE terms will be coded by Medical Dictionary for Regulatory Activities (MedDRA) Version 19.1 and will be presented by system organ class (SOC) and preferred term (PT). Treatment-emergent AEs will be summarized by SOC and PT and by CTCAE toxicity grade. The drug-related AEs, serious adverse events (SAEs) and drug-related SAEs, AEs leading to treatment discontinuation, dose delay and dose modification will be summarized by PT by CTCAE toxicity grade.

Death will be reported in a listing and summarized. A table will be provided for grade 5 AE and the relationship with any study drug.

#### 10.6.1 Adverse Events of Clinical Interest

In addition to general analyses of adverse events, analyses will be conducted on selected AEs of clinical interest. The following are event of clinical interests (ECIs): cardiac events (including atrial fibrillation), anemia, cytopenias, hemorrhage including major hemorrhage, hepatic events, hypertension, infections, interstitial lung disease and pneumonitis, second primary malignancies, and tumor lysis syndrome. Details of ECIs is summarized in the Appendices of this SAP.

AEs of clinical interest are defined in section 14.4 of the appendices.

Subject incidence rates of AEs of clinical interest will be tabulated by treatment cohorts and all-treated population.

Acerta Pharma 

#### 10.6.2 **Laboratory Abnormality**

All of the laboratory tests are performed in central laboratory and/or in local laboratory. Analyses will be performed for laboratory test data collected at baseline and from first exposure to acalabrutinib to 30 days after last dose of acalabrutinib or up to the safety follow-up visit date, whichever is later. Laboratory test for hematology, serum chemistry, and T/B/NK cell count up will be performed in central laboratory with reference range and the results will be reported in standard international units or conventional units when appropriate. Applicable laboratory test results will be graded according to CTCAE Version 4.03 or higher. AMA (American Medical Association (AMA) Manual of Style 10<sup>th</sup> Edition 2017) laboratory values will be applied whenever reference ranges are not available (e.g., local laboratory data).

For selected laboratory test parameters, summary statistics (mean, standard deviation, median, minimum and maximum) will be produced at baseline, post-baseline values from the last visit, minimum and maximum post-baseline values, and changes of these post-baseline values from baseline. Post-baseline toxicity grade greater than baseline grade will be presented in the treatment-emergent laboratory abnormality table. Shift from baseline to the worst grade from first exposure to acalabrutinib to 30 days after last dose of acalabrutinib or up to the safety follow-up visit date, whichever is later, will be provided as shift tables for selected parameters.

To be included in the summary table, a subject must have at least one post-baseline value for the given time point.

#### Lymphocytosis

Lymphocytosis is defined as an elevation in absolute lymphocyte count (ALC) of  $\geq$  50% compared to baseline and a post-baseline assessment  $>5x10^9/L$  (Wang 2013). The number of subjects with at least one occurrence of lymphocytosis will be summarized. For subjects with lymphocytosis, resolution of lymphocytosis is defined as 1) a decrease of ALC value to the baseline level or lower, or 2) a decrease of ALC value that is below  $5x10^9/L$ , whichever occurs first. Duration of lymphocytosis (DOL) is defined as the duration of time from the earliest date on which the ALC value met the lymphocytosis criteria at a post-baseline assessment to the earliest date on which a subsequent ALC value met the resolution criteria.

Acerta Pharma 

DOL = Earliest date of meeting resolution criteria -Earliest date of meeting lymphocytosis criteria + 1.

Subjects who developed lymphocytosis but whose lymphocytosis was not resolved prior to the analysis cutoff date will be censored at the last sample date with non-missing ALC value at or prior to the analysis cutoff date.

Summary statistics will be provided for time to lymphocytosis. KM estimates for DOL will be provided.

#### Hepatitis B Test

Subjects with a history of hepatitis B virus (HBV) infection should be monitored monthly with a quantitative polymerase chain reaction (PCR) test for HBV DNA. Monthly monitoring should last until 12 months after last dose of acalabrutinib. Any subject with a rising viral load (above lower limit of detection) should discontinue study drug and have antiviral therapy instituted and a consultation with a physician with expertise in managing hepatitis B. A listing of subjects with any hepatitis B test will be provided.

## 10.6.3 Vital Signs

Analyses will be performed for vital sign safety data collected at baseline and from first exposure to acalabrutinib to 30 days after last dose of acalabrutinib or up to the safety follow-up visit date, whichever is later. Summary statistics (mean, standard deviation, median, minimum and maximum) will be produced for vital signs at baseline, post-baseline values from the last visit, minimum and maximum post-baseline values, and changes of these post-baseline values from baseline. In addition, blood pressure is graded and the maximum post-baseline grade will be presented. Systolic Blood Pressure is graded by CTCAE as Grade 0 (<= 119 mm Hg), Grade 1 (120-139 mm Hg), Grade 2 (140 – 159 mm Hg), Grade 3 (>= 160 mm Hg). Diastolic Blood Pressure is grade as Grade 0 (<= 79 mm Hg), Grade 1 (80 -89 mm Hg), Grade 2 (90 – 99 mm Hg), Grade 3 (>= 100 mm Hg). In order to be included in the table, a subject must have at least one post-baseline value for the given time point.

#### 10.6.4 **ECOG Performance Score**

Change of ECOG score from baseline to the worst score during the period from first exposure to acalabrutinib to 30 days after last dose of acalabrutinib or up to the safety follow-up visit date, whichever is later will be provided as shift tables.

Acerta Pharma 

#### 10.6.5 **Electrocardiogram**

ECG data are collected at screening. The investigator assessment of clinical significance categorized as normal, abnormal but not clinically significant, and abnormal clinically significant will be summarized. The number of subjects with corrected QT interval (QTc) greater than 480 msec will also be provided. A listing of subjects with abnormal and clinically significant baseline ECG results or QTc> 480 msec will be provided.

## 10.7 Analyses of Efficacy Endpoints

#### 10.7.1 **Definitions**

Study treatment response will be assessed according to response criteria of standardized tumor response and disease progression for MM ([Rajkumar 2011] and [Blade 1998]) including stringent complete response (sCR), complete response (CR), very good partial response (VGPR), partial response (PR), minimal response (MR), stable disease (SD), and disease progression. Overall response data will be summarized as follows:

Overall Response Rate

ORR is defined as the proportion of subjects who achieve a sCR, CR, VGPR, or PR.

Clinical Benefit Rate

Clinical benefit rate (CBR) is defined as the proportion of subjects who achieve a sCR, CR, VGPR, PR, or MR.

Disease Control Rate

Disease control rate (DCR) is defined as the proportion of subjects who achieve a sCR, CR, VGPR, PR, MR, or SD.

Duration of Response (DOR)

DOR is defined as the interval from the first documentation of sCR, CR, VGPR or PR to the first documentation of definitive disease progression or death from any cause. Data from surviving, non-progressing subjects will be censored at the earliest of the time of initiation of anticancer treatment other than the study treatment or the last time that lack of definitive MM progression was objectively documented. Data from subjects who have

Acerta Pharma 

MM progression or die after ≥ 2 consecutive missing tumor assessments will be censored at the last time before the missing assessments that lack of MM progression was objectively documented. The censoring rules for analyses of DOR are summarized in Appendix 14.3.

#### Progression-free Survival (PFS)

PFS is defined as the interval between the date of randomization to any study cohort and the first documentation of objective MM disease progression or death from any cause. Data from surviving, non-progressing subjects will be censored at the earliest of the time of initiation of anticancer treatment other than the study treatment or the last time that lack of MM progression was objectively documented. Subjects who have MM progression or die after ≥ 2 consecutive missing tumor assessments will be censored at the last time that lack of MM progression was objectively documented before the missing assessments. The censoring rules for analyses of PFS are summarized in Appendix 14.3.

#### 10.7.2 **Analysis Methods**

The analysis of ORR, CBR, DCR, and PFS will be conducted on the All-treated Population. The analysis of DOR will be conducted on the subset of the All-treated Population who achieve sCR, CR, VGPR or PR as their best overall response.

ORR, CBR, DCR will be calculated and the corresponding 95% two-sided confidence intervals will be derived. DOR and PFS will be estimated using the Kaplan-Meier (KM) method. KM estimates with 95% CIs will be calculated for event time quartiles, including median. In addition, listings for DOR and PFS will be provided, including the reason for censoring.

#### 11. **DISEASE BIOMARKERS**

The relationship between biological markers in MM cells and response to therapy will not be explored, due to the fact that a very small number of subjects has responded to study treatment.

#### 12. **CHANGES FROM PROTOCOL-SPECIFIED ANALYSES**

There is no major change from protocol-specified analyses.

Acerta Pharma 

#### 13. LITERATURE CITATIONS / REFERENCES

The American Medical Association (AMA) Manual of Style, SI Conversion Calculator,

http://www.amamanualofstyle.com/page/si-conversion-calculator

Anderson KC, Alsina M, Bensinger W, et al. Multiple myeloma, version 1.2013. J Natl Compr Canc Netw 2013;11:11-17.

Bladé J, Samson D, Reece D, et al. Criteria for evaluating disease response and progression in patients with multiple myeloma treated by high-dose therapy and haemopoietic stem cell transplantation. Myeloma Subcommittee of the EBMT. European Group for Blood and Marrow Transplant. Br J Haematol 1998;102:1115-1123.

Cheson BD, Pfistner B, Juweid ME, et al. Revised response criteria for malignant lymphoma. J Clin Oncol 2007; 25:579-586.

Cheson BD, Fisher RI, Barrington SF, et al. Recommendations for initial evaluation, staging, and response assessment of Hodgkin and non-Hodgkin lymphoma: the Lugano classification. J Clin Oncol 2014;32:3059-3067.

Common Terminology Criteria for Adverse Events (CTCAE) Version 4.0, USDHHS, NIH, NCI; publish date May 28, 2009 (v4.03: June 14, 2010).

Rajkumar SV, Harousseau JL, Durie B, et al; International Myeloma Workshop Consensus Panel 1. Consensus recommendations for the uniform reporting of clinical trials: report of the International Myeloma Workshop Consensus Panel 1. Blood. 2011 May 5;117(18):4691-5.

Greipp PR, Miguel JS, Durie BGM, Crowley JJ, Barlogie B, et al; International Staging System for Multiple Myeloma: Journal of Clinical Oncology 2005 23:15, 3412-3420.

Wang ML, Rule S, Martin P, et al. Targeting BTK with ibrutinib in relapsed or refractory mantle-cell lymphoma. N Engl J Med 2013 Aug 8;369(6):507-516.

#### 14. APPENDICES

#### 14.1 Definitions

## 14.1.1 **Study Day**

The study day will be calculated in reference to the date of first dose date. Study Day 1 is defined as the date of first dose of acalabrutinib. For assessments that occur on or after first dose date, study day is defined as (date of assessment – date of first dose + 1). For assessments that occur prior to first dose date, study day is defined as (date of assessment – date of first dose). There is no Study Day 0.

## 14.2 Imputation Rules

## 14.2.1 Partial or Missing Dates

Imputation of partial dates will be made for AE onset and stop dates, start and end dates of concomitant medication, start date of subsequent anticancer therapy, date of initial diagnosis and death date. If dates are completely missing, no imputation will be made. For any partial date with missing year, no imputation will be made.

The general rule for imputation is:

- If only day is missing, then the 15<sup>th</sup> of the month will be used.
- If only year is present, then June 30<sup>th</sup> will be used.

If such imputation date for initial diagnosis is on or after date of first dose, the date of first dose – 1 will be used. If such imputed date for subsequent anticancer therapies is before date of last dose, the date of last dose + 1 will be used.

If the imputed date is for an AE start date and is in the same year and month as the first dose date but before the first dose date, the first dose date will be used, or if the imputed AE start date is after the AE end date, the AE end date will be used. If the imputed date is for an AE start date and is in the same year and month as but after the last dose date + 30 days, the last dose date + 30 days will be used.

If the imputed date is for an AE end date and is after the death date, the date of death will be used, or if the imputed AE end date is before the AE start date, the AE start date will be used.

If death year and month are available but day is missing:

Acerta Pharma 

- If mmyyyy for last contact date = mmyyyy for death date, set death date to the day after the last contact date.
- If mmyyyy for last contact date < mmyyyy for death date, set death date to the first day of the death month.
- If mmyyyy for last contact date > mmyyyy for death date, data error and do not impute.

If both month and day are missing for death date or a death date is totally missing, no imputation is made.

# 14.3 Censoring Rules for Duration of Response and Progression-Free Survival

| Situation | Outcome | Event Description or Censoring Reason | Last Analysis<br>Date |
|---|---|---|---|
| Documented disease progression<br>before initiation of new anticancer<br>therapy or on/before data cutoff<br>date, whichever occurred first, also<br>no more than 1 missing tumor<br>assessments before documented<br>disease progression | Event | Progressive<br>Disease | Earliest date of<br>documented<br>disease<br>progression |
| Death before initiation of new anticancer therapy or on/before data cutoff date, whichever occurred first | Event | Death | Date of Death |
| New anticancer therapy<br>Initiated before data cutoff date and<br>before documented disease<br>progression or death | Censored | New anti-cancer<br>therapy | Date of last<br>adequate tumor<br>assessment prior<br>to initiation of new<br>anticancer<br>therapy |
| New anti-cancer therapy<br>before data cutoff date for subjects<br>without documented disease<br>progression or death | Censored | New anti-cancer<br>therapy | Date of last<br>adequate tumor<br>assessment prior<br>to initiation of new<br>anticancer<br>therapy |
| No documented disease progression, initiation of new anticancer therapy or death on/before data cutoff date | Censored | Data cutoff | Date of last<br>adequate tumor<br>assessment on or<br>before data cutoff<br>date |
| No post-baseline adequate disease assessments | Censored | No post-baseline adequate disease assessments | Date of first dose of study drug |

## 14.4 Events of Clinical Interest

The Events of Clinical Interest (ECIs) have been identified based on preclinical findings, emerging data from clinical studies relating to acalabrutinib, and pharmacological effects

Acerta Pharma 

of approved BTK inhibitor. The AEs selected for dedicated analysis were evaluated using Standardized MedDRA Queries (SMQs), where available, by SOC, or by sponsor defined baskets of MedDRA Adverse Event Grouped Terms.

| Category | Sub- | Definition for SAP | Additional Criteria for Narratives |
|---|---|---|---|
| name | category | | |
| | name | | |
| Cardiac events | | SOC Cardiac disorders | No additional criteria |
| | Atrial | PT Atrial fibrillation | Any |
| | fibrillation | PT Atrial flutter | |
| Cytopenias- | | SMQ Haematopoietic | No additional criteria |
| Anemia | | erytheropenia [narrow + broad] | |
| Cytopenias- | | SMQ Haematopoietic | No additional criteria |
| Leukopenia | | leukopenia [narrow + broad] | |
| | Neutropenia | PT Febrile neutropenia | No additional criteria |
| | | PT Neutropenia | |
| | | PT Neutropenic infection | |
| | | PT Neutropenic sepsis | |
| | | PT Neutrophil count | |
| | | decreased | |
| | | PT Neutrophil percentage | |
| | Other | SMQ Haematopoietic | No additional criteria |
| | Leukopenia | leukopenia [narrow + broad] | |
| | | excluding PTs for neutropenia | |
| | | above | |
| Cytopenias - | | SMQ Haemorrhage terms | No additional criteria |
| Thrombocytop | | (excluding laboratory terms) | |
| enia | | | |
| | Major | As per Acerta definition | Any |
| | Hemorrhage | (Appendences) | |
| Hepatic Events | | SMQ [narrow] Hepatic | PTs of Grade ≥3 as below |
| | | failure, fibrosis and cirrhosis | Alanine aminotransferase |
| | | and other liver damage | abnormal |
| | | related conditions | Alanine aminotransferase |
| | | SMQ [narrow] Liver related | increased |
| | | investigation signs | Aspartate aminotransferase |
| | | SMQ [narrow] Hepatitis, non- | abnormal |
| | | infectious | Aspartate aminotransferase |
| | | | increased |
| | | | Hepatic enzyme abnormal |
| | | | Hepatic enzyme increased |
| | | | Hypertransminasemia |

Acerta Pharma 

| | ı | | |
|---|---|---|---|
| | | | Liver function test abnormal |
| | | | Liver function test increase |
| | | | <ul> <li>Transaminases abnormal</li> </ul> |
| | | | Transaminases increased |
| | | | Subjects who fulfill biochemical Hy's |
| | | | law criteria defined as below: |
| | | | ≥ 3 x ULN AST or |
| | | | ≥ 3 x ULN ALT and |
| | | | ≥ 2 x ULN total bilirubin |
| | | | At the same visit |
| Hypertension | | SMQ Hypertension [narrow] | No additional criteria |
| Infections | | SOC Infections and | No additional criteria |
| | | infestations | |
| Interstitial lung | | SMQ [narrow] Interstitial lung | No additional criteria |
| disease/Pneu | | disease | |
| monitis | | | |
| Second | | SMQ Malignant or | Any |
| primary | | unspecified tumors and | |
| malignancies | | SMQ Myelodysplastic | |
| | | syndrome (narrow), | |
| | | excluding skin (i.e. exclude | |
| | | SMQ Skin neoplasms, | |
| | | malignant and unspecified) | |
| Tumor lysis | | PT Tumor lysis syndrome | Any |
| syndrome | | | |
| | | | ı |

MedDRA version 19.1

- No additional criteria means only SAE, AE leading to study drug discontinuation, and deaths within specified window will be selected for narratives.
- 'Any' means any subject with a PT in the category will be selected for narratives.

Acerta Pharma 